CLINICAL TRIAL: NCT03799380
Title: DRIHNC - Dehydration Reduction in Head & Neck Cancer: Daily Oral Fluid and Electrolyte Maintenance to Prevent Acute Care Clinic and Emergency Department Visits for Patients Receiving Radiation With or Without Chemotherapy/Immunotherapy for Head & Neck and Esophageal Cancer.
Brief Title: DRIHNC - Dehydration Reduction in Head & Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8318
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Dehydration; Head & Neck Cancer; Esophageal Cancer
MeSH Terms: conditions — Dehydration; Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard of Care (Active Comparator): Standard of care nutritional support
  Interventions: Dietary Supplement: Standard of care nutritional support
- Experimental - Gatorade (Experimental): Standard of care nutritional support with the addition of daily Gatorade G2
  Interventions: Dietary Supplement: Gatorade G2

INTERVENTIONS:
Dietary Supplement: Gatorade G2 — Gatorade (G2), 20 oz. bottle, daily through the entire course of radiation therapy (approximately 5-7 weeks)
  Arms: Experimental - Gatorade
Dietary Supplement: Standard of care nutritional support — Standard of care nutritional support
  Arms: Control - Standard of Care

SUMMARY:
The purpose of this study is to decrease the rate of visits to the Emergency Department (ED) and Acute Care Clinics (ACC) for dehydration for head & neck (H&N) and esophageal cancer patients that are given Gatorade while receiving radiation therapy with or without chemotherapy.

DETAILED DESCRIPTION:
Among patients with cancer of the H&N or esophagus, complications related to dehydration are fairly common, and can result in requiring IV fluid support in an ACC setting, ED or even inpatient admission. By instructing participants to drink a reasonable amount of a common electrolyte-rich energy drink from the initiation of treatment through its completion, the hypothesis will be tested that this inexpensive and easily administered preventative strategy can significantly decrease the rate of ACC and ED visits.

The objectives of this study are to decrease the frequency of ACC visits during the course of radiation therapy and decrease the frequency of ED visits during the course of radiation therapy. The study team also seeks to decrease the incidence of orthostatic vital signs during the course of radiation therapy and decrease the number of days of missed treatments due to radiation toxicity during the course of radiation therapy.

In the pilot cohort, participants will be given Gatorade G2 to drink daily during the course of radiation, along with standard of care nutritional support from dietitians. The randomized Phase 2 cohort has two study groups. Group 1 will receive standard of care nutritional support. Group 2 will receive standard of care nutritional support plus the study agent, Gatorade G2.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must have histologically confirmed primary invasive cancer of the H&N (Nasopharynx/Nasal Cavity, Oral cavity, Oropharynx, Larynx, Hypopharynx) or Esophagus.

Histologies: squamous cell carcinoma, adenocarcinoma, adenoid cystic carcinoma, sinonasal undifferentiated carcinoma Stages: Any stage that necessitates radiation therapy (either definitive, neoadjuvant or adjuvant) as per standard practice guidelines (NCCN, ASTRO)

* Subjects must have received no prior radiation therapy to the head, neck, thorax or abdomen in the last 1 year (with the exception of scalp squamous cell or basal cell carcinoma.
* ECOG Performance status 0-2.
* Life expectancy of ≥ 3 months, in the opinion of and as documented by the investigator.
* Subjects must have organ and marrow function based on lab values deemed acceptable to proceed with radiation therapy. No additional or specific lab value cutoffs are required for this protocol given the nature of the intervention. General guidelines are provided below.
* Hemoglobin ≥ 7 g/dl
* Absolute neutrophil count ≥ 500/mcL
* Platelet count ≥ 50,000/mcL
* Total bilirubin within normal institutional limits
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* HIV-positive subjects on combination antiretroviral therapy are eligible.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment.

* Prior radiation therapy to the head, neck, thorax or abdomen in the last year, with the exception of scalp squamous cell or basal cell carcinoma.
* Patients with active, uncontrolled, symptomatic volume overload congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
ACC visits | Up to 11 weeks after start of treatment
  ACC visits during the course of radiation (7 weeks). Participants are followed for 4 weeks after completion of radiation.
ED visits | Up to 11 weeks after start of treatment
  Number of ED visits during the course of radiation (7 weeks). Participants are followed for 4 weeks after completion of radiation.

SECONDARY OUTCOMES:
Incidence of orthostatic vital signs | Up to 11 weeks after start of treatment
  Number of orthostatic vital signs during the course of radiation therapy assessed at weekly visits.
Missed days of radiation +/- chemotherapy/immunotherapy treatment | Up to 7 weeks after start of treatment
  Number of missed days of radiation treatment among H&N and esophageal cancer patients undergoing radiation +/- chemotherapy/immunotherapy during the course of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elisha Fredman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States